CLINICAL TRIAL: NCT06580314
Title: A Phase III Trial of One vs. Two Years of Maintenance Olaparib, With or Without Bevacizumab, in Patients With BRCA1/2 Mutated or Homologous Recombination Deficient (HRD+) Ovarian Cancer Following Response to First Line Platinum-Based Chemotherapy
Brief Title: Testing Olaparib for One or Two Years, With or Without Bevacizumab, to Treat Ovarian Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: NRG Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NRG-GY036; NCI-2024-04335 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NRG-GY036 (Other: NRG Oncology); NRG-GY036 (Other: CTEP); U10CA180868 (NIH)
Record Dates: First submitted 2024-08-28; First posted 2024-08-30 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Fallopian Tube Endometrioid Adenocarcinoma; Fallopian Tube High Grade Serous Adenocarcinoma; FIGO Stage III Ovarian Cancer 2014; FIGO Stage IV Ovarian Cancer 2014; Ovarian Carcinoma; Ovarian High Grade Endometrioid Adenocarcinoma; Ovarian High Grade Serous Adenocarcinoma; Primary Peritoneal Endometrioid Adenocarcinoma; Primary Peritoneal High Grade Serous Adenocarcinoma
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Bevacizumab; Immunoglobulin G; Disulfides; Specimen Handling; Magnetic Resonance Spectroscopy; olaparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm I (olaparib, bevacizumab) (Active Comparator): Patients receive olaparib PO BID on days 1-21 of each cycle. Cycles repeat every 21 days for up to 2 years in the absence of disease progression or unacceptable toxicity. Patients may also receive bevacizumab IV on day 1 of each cycle. Cycles of bevacizumab repeat every 21 days for up to 1 year in the absence of disease progression or unacceptable toxicity. Patients also undergo blood sample collection and CT and/or MRI throughout the study.
  Interventions: Biological: Bevacizumab; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Drug: Olaparib
- Arm II (olaparib, bevacizumab) (Experimental): Patients receive olaparib PO BID on days 1-21 of each cycle. Cycles repeat every 21 days for up to 1 year in the absence of disease progression or unacceptable toxicity. Patients may also receive bevacizumab IV on day 1 of each cycle. Cycles of bevacizumab repeat every 21 days for up to 1 year in the absence of disease progression or unacceptable toxicity. Patients also undergo blood sample collection and CT and/or MRI throughout the study.
  Interventions: Biological: Bevacizumab; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Drug: Olaparib

INTERVENTIONS:
Biological: Bevacizumab — Given IV
  Other Names: ABP 215; ABP-215; ABP215; Alymsys; Anti-VEGF; Anti-VEGF Humanized Monoclonal Antibody; Anti-VEGF Monoclonal Antibody SIBP04; Anti-VEGF rhuMAb; Avastin; Avzivi; Aybintio; BAT 1706; BAT-1706; BAT1706; BAT1706 Biosimilar; Bevacizumab awwb; Bevacizumab Biosimilar ABP 215; Bevacizumab Biosimilar BAT1706; Bevacizumab Biosimilar BEVZ92; Bevacizumab Biosimilar BI 695502; Bevacizumab Biosimilar CBT 124; Bevacizumab Biosimilar CT-P16; Bevacizumab Biosimilar FKB238; Bevacizumab Biosimilar GB-222; Bevacizumab Biosimilar HD204; Bevacizumab Biosimilar HLX04; Bevacizumab Biosimilar IBI305; Bevacizumab Biosimilar LY01008; Bevacizumab Biosimilar MB02; Bevacizumab Biosimilar MIL60; Bevacizumab Biosimilar Mvasi; Bevacizumab Biosimilar MYL-1402O; Bevacizumab Biosimilar QL 1101; Bevacizumab Biosimilar QL1101; Bevacizumab Biosimilar RPH-001; Bevacizumab Biosimilar SCT501; Bevacizumab Biosimilar Zirabev; Bevacizumab-adcd; Bevacizumab-awwb; Bevacizumab-aybi; Bevacizumab-bvzr; Bevacizumab-equi; Bevacizumab-maly; Bevacizumab-onbe; Bevacizumab-tnjn; BP102; BP102 Biosimilar; CT P16; CT-P16; CTP16; Equidacent; FKB 238; FKB-238; FKB238; HD204; Immunoglobulin G1 (Human-Mouse Monoclonal rhuMab-VEGF Gamma-Chain Anti-Human Vascular Endothelial Growth Factor), Disulfide With Human-Mouse Monoclonal rhuMab-VEGF Light Chain, Dimer; MB 02; MB-02; MB02; Mvasi; MYL-1402O; Onbevzi; Oyavas; PF 06439535; PF-06439535; PF06439535; QL1101; Recombinant Humanized Anti-VEGF Monoclonal Antibody; rhuMab-VEGF; SCT501; SIBP 04; SIBP-04; SIBP04; Vegzelma; Zirabev
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Drug: Olaparib — Given PO
  Other Names: AZD 2281; AZD-2281; AZD2281; KU 0059436; KU-0059436; KU0059436; Lynparza; Olanib; Olaparix; PARP Inhibitor AZD2281

SUMMARY:
This phase III trial compares the effect of olaparib for one year versus two years, with or without bevacizumab, for the treatment of BRCA 1/2 mutated or homologous recombination deficient stage III or IV ovarian cancer. Olaparib is a polyadenosine 5'-diphosphoribose polymerase (PARP) enzyme inhibitor and may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Bevacizumab is in a class of medications called antiangiogenic agents. It works by stopping the formation of blood vessels that bring oxygen and nutrients to tumor. This may slow the growth and spread of tumor. Giving olaparib for one year with or without bevacizumab may be effective in treating patients with BRCA 1/2 mutated or homologous recombination deficient stage III or IV ovarian cancer, when compared to two years of olaparib.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine investigator assessed progression-free survival using Response Evaluation Criteria in Solid Tumors (RECIST) version (v)1.1 (non-inferiority) for one versus (vs.) two years of maintenance olaparib.

SECONDARY OBJECTIVES:

I. To evaluate overall survival (OS360) in the modified intent to treat (ITT) population, with time at risk for progression/death starting 360 days after randomization.

II. To evaluate progression-free survival (PFS), PFS2 and overall survival (OS) in the ITT population.

III. To evaluate PFS, PFS2, and OS in the as-treated population. IV. To evaluate toxicity, including rates of myelodysplastic syndrome (MDS), acute myeloid leukemia (AML), and other secondary malignancies, in the safety population.

EXPLORATORY OBJECTIVE:

I. To evaluate the moderating effect of physician-choice bevacizumab (as stratified) on randomized treatment effect estimates.

TRANSLATIONAL OBJECTIVES:

I. To assess BRCA reversion mutations in circulating tumor deoxyribonucleic acid (ctDNA) as a predictor of poor response in the BRCA mutated (BRCAm) population.

II. To correlate a combined assay assessing quantitative BRCA1 and RAD51C promoter methylation and pathogenic variants in core homologous recombination repair (HRR) genes with clinical homologous recombination deficiency (HRD) testing and outcomes in the BRCA wildtype (BRCAwt) population.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I (REFERENCE): Patients receive olaparib orally (PO) twice daily (BID) on days 1-21 of each cycle. Cycles repeat every 21 days for up to 2 years in the absence of disease progression or unacceptable toxicity. Patients may also receive bevacizumab IV on day 1 of each cycle. Cycles of bevacizumab repeat every 21 days for up to 1 year in the absence of disease progression or unacceptable toxicity. Patients also undergo blood sample collection and computed tomography (CT) and/or magnetic resonance imaging (MRI) throughout the study.

ARM II (EXPERIMENTAL): Patients receive olaparib PO BID on days 1-21 of each cycle. Cycles repeat every 21 days for up to 1 year in the absence of disease progression or unacceptable toxicity. Patients may also receive bevacizumab IV on day 1 of each cycle. Cycles of bevacizumab repeat every 21 days for up to 1 year in the absence of disease progression or unacceptable toxicity. Patients also undergo blood sample collection and CT and/or MRI throughout the study.

After completion of study treatment, patients are followed up every 3 months for 2 years, then every 6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients with newly diagnosed, pathologically confirmed, Federation of Gynecology and Obstetrics (FIGO) stage III or IV ovarian cancer of the following types:

  * High grade serous
  * High grade endometrioid, and/or
  * Other epithelial ovarian cancer with BRCA1/2 deleterious alteration (germline or somatic)
  * Submission of pathology report is required
  * Ovarian cancer = ovarian, fallopian, or primary peritoneal cancer
* Patients must have:

  * Documented variant (tumor or germline) in BRCA1 or BRCA2 that is predicted to be pathogenic or suspected pathogenic (deleterious alteration)

    * Submission of testing report is required. OR
  * BRCA 1/2 wildtype AND known HRD deficient tumor determined by any commercial or academic, Clinical Laboratory Improvement Act (CLIA)-certified laboratory (e.g., Myriad MyChoice©)

    * Submission of testing report is required
* Patient must have undergone cytoreductive surgery (primary or interval)
* Patients must have completed first line platinum-based therapy prior to registration:

  * Platinum based chemotherapy course must have consisted of a minimum of 4 treatment cycles and a maximum of 9, although it is strongly recommended that patients receive at least 6 cycles unless medically contraindicated

    * For those receiving less than 6 cycles of platinum-based therapy, the reason for this must be documented and could include hematologic toxicity or non-hematologic toxicities directly related to therapy
  * Intravenous, intraperitoneal, or neoadjuvant platinum-based chemotherapy is allowed; for weekly therapy, three weeks are considered one cycle
  * Patients must not have received an investigational agent during their first line course of chemotherapy
* Patients must have, in the opinion of the investigator, no clinical evidence of disease progression following completion of this chemotherapy course (partial or complete response to platinum-based chemotherapy)
* Patients with treated brain metastases are eligible if follow up brain imaging after central nervous system (CNS) directed therapy shows no evidence of progression following completion of this chemotherapy course (partial or complete response to platinum-based chemotherapy)
* Patients must be randomized at least 3 weeks and no more than 12 weeks after their last dose of chemotherapy (last dose is the day of the last infusion of platinum agent)
* No previous treatment with a PARP inhibitor, including olaparib, niraparib, and rucaparib
* Age ≥ 18
* Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 2
* Not pregnant and not nursing
* Absolute neutrophil count (ANC) ≥ 1,500 cells/mm^3
* Platelets ≥ 100,000 cells/mm^3
* Hemoglobin ≥ 9 g/dl
* Creatinine clearance (CrCL) of > 30 mL/min by the Cockcroft-Gault formula
* Total bilirubin ≤ 1.5 x institutional upper limit of normal (ULN) (patients with known Gilbert's disease who have bilirubin level ≤ 3 x institutional ULN may be enrolled)
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3 x institutional ULN
* Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, patients should be class 2B or better
* No active infection requiring parental antibiotic(s)
* No current evidence of intra-abdominal abscess, abdominal/pelvic fistula (not diverted), gastrointestinal perforation, gastrointestinal (GI) obstruction, and/or need for drainage nasogastric or gastrostomy tube
* No current inability to swallow orally administered medication
* No history of myelodysplastic syndrome and/or acute myeloid leukemia
* No history of allogeneic bone marrow transplant
* No concomitant use of strong or moderate CYP3A inducers
* No known hypersensitivity to olaparib or any of the excipients of the product

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 880 (Estimated)
Dates: Start 2025-03-12 (Actual); Primary Completion 2034-12-31 (Estimated); Study Completion 2034-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) at least 360 days after randomization (PFS360) | From completing 360 days of maintenance therapy to disease progression (per Response Evaluation Criteria in Solid Tumors [RECIST] version [v]1.1) or death, whichever occurs first, assessed up to 5 years
  PFS will be tested using a one-sided, alpha = 0.05 level logrank test. Treatment hazard ratios and their 90% confidence intervals will be estimated using a Cox proportional hazards model specified with a main effect for the randomized treatment assignment and stratified using the stratification factors applied at randomization.

SECONDARY OUTCOMES:
Overall survival (OS) 360 | From 360 days after randomization to death from any cause, assessed up to 5 years
  This endpoint will be supported by the modified intent to treat (ITT) population, which excludes progressions, deaths or withdrawals within 359 days of randomization. Will be summarized using treatment hazard ratio estimates (90% confidence intervals). These estimates will be obtained from outcome-specific Cox-regression models specified with main effects for the randomized treatment and stratified by the factors included in the randomization. OS distributions will be summarized using methods developed by Kaplan-Meier.
PFS | From randomization to progression or death, whichever occurs first, or date of the last computed tomography scan if neither progression nor death has occurred, assessed up to 5 years
  Will be analyzed in the ITT population and serve as a sensitivity analysis for the primary endpoint. Will be summarized using treatment hazard ratio estimates (90% confidence intervals). These estimates will be obtained from outcome-specific Cox-regression models specified with main effects for the randomized treatment and stratified by the factors included in the randomization. PFS distributions will be summarized using methods developed by Kaplan-Meier.
PFS2 | From randomization to objective tumor progression on next-line treatment or death, assessed up to 5 years
  PFS2 may be identified by objective radiological progression using Response Evaluation Criteria in Solid Tumors version (v)1.1., symptomatic deterioration or death. PFS2 will be summarized using treatment hazard ratio estimates (90% confidence intervals). These estimates will be obtained from outcome-specific Cox-regression models specified with main effects for the randomized treatment and stratified by the factors included in the randomization. PFS2 distributions will be summarized using methods developed by Kaplan-Meier.
OS | From randomization to death, assessed up to 5 years
  OS will be summarized using treatment hazard ratio estimates (90% confidence intervals). These estimates will be obtained from outcome-specific Cox-regression models specified with main effects for the randomized treatment and stratified by the factors included in the randomization. OS distributions will be summarized using methods developed by Kaplan-Meier.
Incidence of adverse events (AEs) | Up to 30 days after last dose of study treatment
  Safety and tolerability will be graded using Common Terminology Criteria for Adverse Events v 5.0. AEs will be summarized by system organ class and preferred term according to the maximum grade observed for each patient.

OTHER OUTCOMES:
Effect of bevacizumab on PFS | Up to 5 years
  The estimates will be obtained from outcome-specific Cox regression models specified with main effects for the assigned treatment arm, physician-choice bevacizumab and the interaction term. The overall effect of bevacizumab will be described by the score test p value for the interaction term. Descriptively, the bevacizumab effect will be summarized using the randomized treatment hazard ratio estimates (95% confidence intervals) within the bevacizumab and no-bevacizumab subgroups (as stratified). PFS outcome distributions will further be described using methods developed by Kaplan-Meier.
Effect of bevacizumab on OS | Up to 5 years
  The estimates will be obtained from outcome-specific Cox regression models specified with main effects for the assigned treatment arm, physician-choice bevacizumab and the interaction term. The overall effect of bevacizumab will be described by the score test p value for the interaction term. Descriptively, the bevacizumab effect will be summarized using the randomized treatment hazard ratio estimates (95% confidence intervals) within the bevacizumab and no-bevacizumab subgroups (as stratified). OS outcome distributions will further be described using methods developed by Kaplan-Meier.
Effect of bevacizumab on PFS2 | Up to 5 years
  The estimates will be obtained from outcome-specific Cox regression models specified with main effects for the assigned treatment arm, physician-choice bevacizumab and the interaction term. The overall effect of bevacizumab will be described by the score test p value for the interaction term. Descriptively, the bevacizumab effect will be summarized using the randomized treatment hazard ratio estimates (95% confidence intervals) within the bevacizumab and no-bevacizumab subgroups (as stratified). PFS2 outcome distributions will further be described using methods developed by Kaplan-Meier.

CONTACTS AND LOCATIONS:
Overall Officials: Ying Liu, Principal Investigator — NRG Oncology
Locations (672):
- United States (654):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Anchorage Associates in Radiation Medicine, Anchorage, Alaska
  - Alaska Breast Care and Surgery LLC, Anchorage, Alaska
  - Alaska Oncology and Hematology LLC, Anchorage, Alaska
  - Alaska Women's Cancer Care, Anchorage, Alaska
  - Katmai Oncology Group, Anchorage, Alaska
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Cancer Center at Saint Joseph's, Phoenix, Arizona
  - Mayo Clinic Hospital in Arizona, Phoenix, Arizona
  - Highlands Oncology Group - Fayetteville, Fayetteville, Arkansas
  - Mercy Hospital Fort Smith, Fort Smith, Arkansas
  - CARTI Cancer Center, Little Rock, Arkansas
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Highlands Oncology Group - Rogers, Rogers, Arkansas
  - Highlands Oncology Group, Springdale, Arkansas
  - Kaiser Permanente-Deer Valley Medical Center, Antioch, California
  - Mission Hope Medical Oncology - Arroyo Grande, Arroyo Grande, California
  - Sutter Auburn Faith Hospital, Auburn, California
  - Sutter Cancer Centers Radiation Oncology Services-Auburn, Auburn, California
  - Kaiser Permanente-Bellflower, Bellflower, California
  - Alta Bates Summit Medical Center-Herrick Campus, Berkeley, California
  - Tower Cancer Research Foundation, Beverly Hills, California
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - Mills-Peninsula Medical Center, Burlingame, California
  - Sutter Cancer Centers Radiation Oncology Services-Cameron Park, Cameron Park, California
  - Mercy Cancer Center - Carmichael, Carmichael, California
  - Mercy San Juan Medical Center, Carmichael, California
  - Eden Hospital Medical Center, Castro Valley, California
  - Sutter Davis Hospital, Davis, California
  - Kaiser Permanente Dublin, Dublin, California
  - Mercy Cancer Center - Elk Grove, Elk Grove, California
  - Stanford Cancer Center Emeryville, Emeryville, California
  - Kaiser Permanente-Fremont, Fremont, California
  - Palo Alto Medical Foundation-Fremont, Fremont, California
  - Fresno Cancer Center, Fresno, California
  - Kaiser Permanente Fresno Orchard Plaza, Fresno, California
  - Kaiser Permanente-Fresno, Fresno, California
  - Kaiser Permanente South Bay, Harbor City, California
  - Kaiser Permanente-Irvine, Irvine, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Kaiser Permanente West Los Angeles, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Mercy Cancer Center, Merced, California
  - Memorial Medical Center, Modesto, California
  - Kaiser Permanente- Modesto MOB II, Modesto, California
  - Kaiser Permanente-Modesto, Modesto, California
  - Palo Alto Medical Foundation-Camino Division, Mountain View, California
  - Palo Alto Medical Foundation-Gynecologic Oncology, Mountain View, California
  - Providence Queen of The Valley, Napa, California
  - Sutter Cancer Research Consortium, Novato, California
  - Kaiser Permanente Oakland-Broadway, Oakland, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Palo Alto Medical Foundation Health Care, Palo Alto, California
  - Stanford Cancer Institute Palo Alto, Palo Alto, California
  - Kaiser Permanente - Panorama City, Panorama City, California
  - Huntington Memorial Hospital, Pasadena, California
  - Kaiser Permanente-Rancho Cordova Cancer Center, Rancho Cordova, California
  - Kaiser Permanente- Marshall Medical Offices, Redwood City, California
  - Kaiser Permanente-Richmond, Richmond, California
  - Kaiser Permanente-Riverside, Riverside, California
  - Mercy Cancer Center - Rocklin, Rocklin, California
  - Rohnert Park Cancer Center, Rohnert Park, California
  - Kaiser Permanente-Roseville, Roseville, California
  - Sutter Cancer Centers Radiation Oncology Services-Roseville, Roseville, California
  - Sutter Roseville Medical Center, Roseville, California
  - The Permanente Medical Group-Roseville Radiation Oncology, Roseville, California
  - Kaiser Permanente Downtown Commons, Sacramento, California
  - Mercy Cancer Center - Sacramento, Sacramento, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - Kaiser Permanente-South Sacramento, Sacramento, California
  - South Sacramento Cancer Center, Sacramento, California
  - Kaiser Permanente-San Diego Zion, San Diego, California
  - California Pacific Medical Center-Pacific Campus, San Francisco, California
  - Kaiser Permanente-San Francisco, San Francisco, California
  - Kaiser Permanente-Santa Teresa-San Jose, San Jose, California
  - Stanford Cancer Center South Bay, San Jose, California
  - Kaiser Permanente San Leandro, San Leandro, California
  - Pacific Central Coast Health Center-San Luis Obispo, San Luis Obispo, California
  - Kaiser Permanente-San Marcos, San Marcos, California
  - Mills Health Center, San Mateo, California
  - Kaiser San Rafael-Gallinas, San Rafael, California
  - Ridley-Tree Cancer Center, Santa Barbara, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Palo Alto Medical Foundation-Santa Cruz, Santa Cruz, California
  - Santa Cruz Radiation Oncology Medical Group, Santa Cruz, California
  - Mission Hope Medical Oncology - Santa Maria, Santa Maria, California
  - Kaiser Permanente-Santa Rosa, Santa Rosa, California
  - Providence Medical Foundation - Santa Rosa, Santa Rosa, California
  - Sutter Pacific Medical Foundation, Santa Rosa, California
  - Providence Santa Rosa Memorial Hospital, Santa Rosa, California
  - Kaiser Permanente Cancer Treatment Center, South San Francisco, California
  - Kaiser Permanente-South San Francisco, South San Francisco, California
  - Saint Joseph's Medical Center, Stockton, California
  - Kaiser Permanente-Stockton, Stockton, California
  - Palo Alto Medical Foundation-Sunnyvale, Sunnyvale, California
  - Torrance Memorial Physician Network - Cancer Care, Torrance, California
  - Kaiser Permanente Medical Center-Vacaville, Vacaville, California
  - Kaiser Permanente-Vallejo, Vallejo, California
  - Sutter Solano Medical Center/Cancer Center, Vallejo, California
  - Kaiser Permanente-Walnut Creek, Walnut Creek, California
  - John Muir Medical Center-Walnut Creek, Walnut Creek, California
  - Woodland Memorial Hospital, Woodland, California
  - Kaiser Permanente-Woodland Hills, Woodland Hills, California
  - UCHealth University of Colorado Hospital, Aurora, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers-Penrose, Colorado Springs, Colorado
  - UCHealth Memorial Hospital Central, Colorado Springs, Colorado
  - Memorial Hospital North, Colorado Springs, Colorado
  - Saint Francis Cancer Center, Colorado Springs, Colorado
  - UCHealth - Cherry Creek, Denver, Colorado
  - CommonSpirit Cancer Center Mercy, Durango, Colorado
  - Mercy Medical Center, Durango, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Cancer Care and Hematology-Fort Collins, Fort Collins, Colorado
  - UCHealth Greeley Hospital, Greeley, Colorado
  - UCHealth Highlands Ranch Hospital, Highlands Ranch, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - Medical Center of the Rockies, Loveland, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - Saint Anthony North Hospital, Westminster, Colorado
  - Danbury Hospital, Danbury, Connecticut
  - Smilow Cancer Hospital Care Center-Fairfield, Fairfield, Connecticut
  - Smilow Cancer Hospital Care Center at Greenwich, Greenwich, Connecticut
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - Smilow Cancer Center/Yale-New Haven Hospital, New Haven, Connecticut
  - Yale University, New Haven, Connecticut
  - Norwalk Hospital, Norwalk, Connecticut
  - Smilow Cancer Hospital Care Center at Long Ridge, Stamford, Connecticut
  - Smilow Cancer Hospital Care Center-Trumbull, Trumbull, Connecticut
  - Smilow Cancer Hospital-Waterbury Care Center, Waterbury, Connecticut
  - Smilow Cancer Hospital Care Center - Waterford, Waterford, Connecticut
  - Beebe Medical Center, Lewes, Delaware
  - Beebe South Coastal Health Campus, Millville, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - Christiana Care Health System-Wilmington Hospital, Wilmington, Delaware
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - Broward Health Medical Center, Fort Lauderdale, Florida
  - UF Health Cancer Institute - Gainesville, Gainesville, Florida
  - Orlando Health Cancer Institute - Lake Mary, Lake Mary, Florida
  - Health Central, Ocoee, Florida
  - Orlando Health Cancer Institute, Orlando, Florida
  - Sacred Heart Hospital, Pensacola, Florida
  - University Cancer and Blood Center LLC, Athens, Georgia
  - Grady Health System, Atlanta, Georgia
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia
  - Northside Hospital, Atlanta, Georgia
  - Augusta University Medical Center, Augusta, Georgia
  - Emory Decatur Hospital, Decatur, Georgia
  - Hawaii Cancer Care Inc - Waterfront Plaza, Honolulu, Hawaii
  - Queen's Cancer Cenrer - POB I, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Kuakini Medical Center, Honolulu, Hawaii
  - Queen's Cancer Center - Kuakini, Honolulu, Hawaii
  - The Cancer Center of Hawaii-Liliha, Honolulu, Hawaii
  - Kaiser Permanente Moanalua Medical Center, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Wilcox Memorial Hospital and Kauai Medical Clinic, Lihue, Hawaii
  - Hawaii Cancer Care - Westridge, ‘Aiea, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - Queen's Cancer Center - Pearlridge, ‘Aiea, Hawaii
  - The Cancer Center of Hawaii-Pali Momi, ‘Aiea, Hawaii
  - The Queen's Medical Center - West Oahu, ‘Ewa Beach, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Kootenai Health - Coeur d'Alene, Coeur d'Alene, Idaho
  - Saint Luke's Cancer Institute - Fruitland, Fruitland, Idaho
  - Idaho Urologic Institute-Meridian, Meridian, Idaho
  - Saint Luke's Cancer Institute - Meridian, Meridian, Idaho
  - Saint Alphonsus Cancer Care Center-Nampa, Nampa, Idaho
  - Saint Luke's Cancer Institute - Nampa, Nampa, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Kootenai Clinic Cancer Services - Sandpoint, Sandpoint, Idaho
  - Saint Luke's Cancer Institute - Twin Falls, Twin Falls, Idaho
  - OSF Saint Anthony's Health Center, Alton, Illinois
  - Rush-Copley Medical Center, Aurora, Illinois
  - Advocate Outpatient Center - Aurora, Aurora, Illinois
  - Advocate Good Shepherd Hospital, Barrington, Illinois
  - Carle BroMenn Outpatient Center, Bloomington, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Memorial Hospital of Carbondale, Carbondale, Illinois
  - SIH Cancer Institute, Carterville, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Saint Mary's Hospital, Centralia, Illinois
  - John H Stroger Jr Hospital of Cook County, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Advocate Illinois Masonic Medical Center, Chicago, Illinois
  - AMG Crystal Lake - Oncology, Crystal Lake, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Illinois CancerCare-Dixon, Dixon, Illinois
  - Advocate Good Samaritan Hospital, Downers Grove, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Advocate Sherman Hospital, Elgin, Illinois
  - Elmhurst Memorial Hospital, Elmhurst, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - Advocate South Suburban Hospital, Hazel Crest, Illinois
  - UChicago Medicine AdventHealth Cancer Institute Hinsdale, Hinsdale, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - AMG Libertyville - Oncology, Libertyville, Illinois
  - Condell Memorial Hospital, Libertyville, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - SSM Health Good Samaritan, Mount Vernon, Illinois
  - Edward Hospital/Cancer Center, Naperville, Illinois
  - UC Comprehensive Cancer Center at Silver Cross, New Lenox, Illinois
  - Carle BroMenn Medical Center, Normal, Illinois
  - Carle Cancer Institute Normal, Normal, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - HSHS Saint Elizabeth's Hospital, O'Fallon, Illinois
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - Advocate Outpatient Center - Oak Lawn, Oak Lawn, Illinois
  - University of Chicago Medicine-Orland Park, Orland Park, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Advocate High Tech Medical Park, Palos Heights, Illinois
  - Advocate Lutheran General Hospital, Park Ridge, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Edward Hospital/Cancer Center?Plainfield, Plainfield, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - UW Health Carbone Cancer Center Rockford, Rockford, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Illinois CancerCare - Washington, Washington, Illinois
  - Rush-Copley Healthcare Center, Yorkville, Illinois
  - IU Health North Hospital, Carmel, Indiana
  - Northwest Cancer Center - Main Campus, Crown Point, Indiana
  - UChicago Medicine Northwest Indiana, Crown Point, Indiana
  - Northwest Oncology LLC, Dyer, Indiana
  - Parkview Regional Medical Center, Fort Wayne, Indiana
  - Goshen Center for Cancer Care, Goshen, Indiana
  - Northwest Cancer Center - Hobart, Hobart, Indiana
  - Saint Mary Medical Center, Hobart, Indiana
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Sidney and Lois Eskenazi Hospital, Indianapolis, Indiana
  - Ascension Saint Vincent Indianapolis Hospital, Indianapolis, Indiana
  - Saint Catherine Hospital, Indianapolis, Indiana
  - The Community Hospital, Munster, Indiana
  - Women's Diagnostic Center - Munster, Munster, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Northwest Cancer Center - Valparaiso, Valparaiso, Indiana
  - Mary Greeley Medical Center, Ames, Iowa
  - McFarland Clinic - Ames, Ames, Iowa
  - McFarland Clinic - Boone, Boone, Iowa
  - Mercy Hospital, Cedar Rapids, Iowa
  - Oncology Associates at Mercy Medical Center, Cedar Rapids, Iowa
  - Heartland Oncology and Hematology LLP, Council Bluffs, Iowa
  - Methodist Jennie Edmundson Hospital, Council Bluffs, Iowa
  - Nebraska Cancer Specialists/Oncology Hematology West PC - MEJ, Council Bluffs, Iowa
  - McFarland Clinic - Trinity Cancer Center, Fort Dodge, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - McFarland Clinic - Jefferson, Jefferson, Iowa
  - McFarland Clinic - Marshalltown, Marshalltown, Iowa
  - Central Care Cancer Center - Garden City, Garden City, Kansas
  - Central Care Cancer Center - Great Bend, Great Bend, Kansas
  - Mercy Hospital Pittsburg, Pittsburg, Kansas
  - Flaget Memorial Hospital, Bardstown, Kentucky
  - Baptist Health Corbin, Corbin, Kentucky
  - Commonwealth Cancer Center-Corbin, Corbin, Kentucky
  - Baptist Health Lexington, Lexington, Kentucky
  - Saint Joseph Hospital, Lexington, Kentucky
  - Saint Joseph Radiation Oncology Resource Center, Lexington, Kentucky
  - Saint Joseph Hospital East, Lexington, Kentucky
  - Saint Joseph London, London, Kentucky
  - The James Graham Brown Cancer Center at University of Louisville, Louisville, Kentucky
  - Baptist Health Louisville, Louisville, Kentucky
  - UofL Health Medical Center Northeast, Louisville, Kentucky
  - Saint Joseph Mount Sterling, Mount Sterling, Kentucky
  - Baptist Health Paducah, Paducah, Kentucky
  - LSU Health Baton Rouge-North Clinic, Baton Rouge, Louisiana
  - Our Lady of the Lake Physician Group, Baton Rouge, Louisiana
  - Our Lady of The Lake, Baton Rouge, Louisiana
  - Our Lady of the Lake Medical Oncology, Baton Rouge, Louisiana
  - West Jefferson Medical Center, Marrero, Louisiana
  - East Jefferson General Hospital, Metairie, Louisiana
  - LSU Healthcare Network / Metairie Multi-Specialty Clinic, Metairie, Louisiana
  - University Medical Center New Orleans, New Orleans, Louisiana
  - Ochsner Baptist Medical Center, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - MaineHealth Maine Medical Center- Scarborough, Scarborough, Maine
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Christiana Care - Union Hospital, Elkton, Maryland
  - Baystate Medical Center, Springfield, Massachusetts
  - MyMichigan Medical Center Gratiot, Alma, Michigan
  - MyMichigan Medical Center Alpena, Alpena, Michigan
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - University of Michigan Rogel Cancer Center, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Brighton, Brighton, Michigan
  - Trinity Health Medical Center - Brighton, Brighton, Michigan
  - University of Michigan - Brighton Center for Specialty Care, Brighton, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Canton, Canton, Michigan
  - Trinity Health Medical Center - Canton, Canton, Michigan
  - Chelsea Hospital, Chelsea, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Chelsea Hospital, Chelsea, Michigan
  - Hematology Oncology Consultants-Clarkston, Clarkston, Michigan
  - Newland Medical Associates-Clarkston, Clarkston, Michigan
  - Henry Ford Health Saint John Hospital, Detroit, Michigan
  - Henry Ford River District Hospital, East China Township, Michigan
  - OSF Saint Francis Hospital and Medical Group, Escanaba, Michigan
  - Cancer Hematology Centers - Flint, Flint, Michigan
  - Genesee Hematology Oncology PC, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - MyMichigan Medical Center Gladwin, Gladwin, Michigan
  - Corewell Health Grand Rapids Hospitals - Butterworth Hospital, Grand Rapids, Michigan
  - Corewell Health Grand Rapids Hospitals - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - Trinity Health Grand Rapids Hospital, Grand Rapids, Michigan
  - Henry Ford Saint John Hospital - Academic, Grosse Pointe Woods, Michigan
  - Henry Ford Saint John Hospital - Breast, Grosse Pointe Woods, Michigan
  - Henry Ford Saint John Hospital - Van Elslander, Grosse Pointe Woods, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Beacon Kalamazoo Cancer Center, Kalamazoo, Michigan
  - Beacon Kalamazoo, Kalamazoo, Michigan
  - University of Michigan Health - Sparrow Lansing, Lansing, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Henry Ford Saint John Hospital - Macomb Medical, Macomb, Michigan
  - Henry Ford Warren Hospital - Breast Macomb, Macomb, Michigan
  - MyMichigan Medical Center Midland, Midland, Michigan
  - MyMichigan Medical Center Mount Pleasant, Mount Pleasant, Michigan
  - Trinity Health Muskegon Hospital, Muskegon, Michigan
  - Corewell Health Lakeland Hospitals - Niles Hospital, Niles, Michigan
  - Cancer and Hematology Centers of Western Michigan - Norton Shores, Norton Shores, Michigan
  - Hope Cancer Center, Pontiac, Michigan
  - Michigan Healthcare Professionals Pontiac, Pontiac, Michigan
  - Newland Medical Associates-Pontiac, Pontiac, Michigan
  - Trinity Health Saint Joseph Mercy Oakland Hospital, Pontiac, Michigan
  - Corewell Health Reed City Hospital, Reed City, Michigan
  - MyMichigan Medical Center Saginaw, Saginaw, Michigan
  - Corewell Health Lakeland Hospitals - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Corewell Health Lakeland Hospitals - Saint Joseph Hospital, Saint Joseph, Michigan
  - MyMichigan Medical Center Tawas, Tawas City, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Henry Ford Health Warren Hospital, Warren, Michigan
  - Henry Ford Madison Heights Hospital - Breast, Warren, Michigan
  - Henry Ford Warren Hospital - GLCMS, Warren, Michigan
  - University of Michigan Health - West, Wyoming, Michigan
  - Huron Gastroenterology PC, Ypsilanti, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology Ann Arbor Campus, Ypsilanti, Michigan
  - Riverwood Healthcare Center, Aitkin, Minnesota
  - Essentia Health - Baxter Clinic, Baxter, Minnesota
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Essentia Health Saint Joseph's Medical Center, Brainerd, Minnesota
  - Minnesota Oncology - Burnsville, Burnsville, Minnesota
  - Cambridge Medical Center, Cambridge, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Essentia Health - Saint Joseph's Crosslake Clinic, Crosslake, Minnesota
  - Essentia Health - Deer River Clinic, Deer River, Minnesota
  - Essentia Health Saint Mary's - Detroit Lakes Clinic, Detroit Lakes, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Essentia Health Saint Mary's Medical Center, Duluth, Minnesota
  - Miller-Dwan Hospital, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Essentia Health - Ely Clinic, Ely, Minnesota
  - Essentia Health - Fosston, Fosston, Minnesota
  - Essentia Health Hibbing Clinic, Hibbing, Minnesota
  - Essentia Health - International Falls Clinic, International Falls, Minnesota
  - Fairview Clinics and Surgery Center Maple Grove, Maple Grove, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Avera Cancer Institute at Marshall, Marshall, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Health Partners Inc, Minneapolis, Minnesota
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - Monticello Cancer Center, Monticello, Minnesota
  - Essentia Health - Moose Lake Clinic, Moose Lake, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - Essentia Health - Park Rapids, Park Rapids, Minnesota
  - Essentia Health - Saint Joseph's Pequot Lakes Clinic, Pequot Lakes, Minnesota
  - Essentia Health - Saint Joseph's Pine River Clinic, Pine River, Minnesota
  - Fairview Northland Medical Center, Princeton, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Essentia Health Sandstone, Sandstone, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Essentia Health - Saint Joseph's Staples Clinic, Staples, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Essentia Health Virginia Clinic, Virginia, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Fairview Lakes Medical Center, Wyoming, Minnesota
  - Mercy Oncology and Hematology - Clayton-Clarkson, Ballwin, Missouri
  - Central Care Cancer Center - Bolivar, Bolivar, Missouri
  - Cox Cancer Center Branson, Branson, Missouri
  - Mercy Cancer Center - Cape Girardeau, Cape Girardeau, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - MU Health - University Hospital/Ellis Fischel Cancer Center, Columbia, Missouri
  - Parkland Health Center - Farmington, Farmington, Missouri
  - Freeman Health System, Joplin, Missouri
  - Mercy Hospital Joplin, Joplin, Missouri
  - Lake Regional Hospital, Osage Beach, Missouri
  - Mercy Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Phelps Health Delbert Day Cancer Institute, Rolla, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Mercy Infusion Center - Chippewa, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital South, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - BJC Outpatient Center at Sunset Hills, Sunset Hills, Missouri
  - Mercy Hospital Washington, Washington, Missouri
  - Community Hospital of Anaconda, Anaconda, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Saint Vincent Frontier Cancer Center, Billings, Montana
  - Intermountain Health West End Clinic, Billings, Montana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Hi-Line Sletten Cancer Center, Havre, Montana
  - Logan Health Medical Center, Kalispell, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Community Medical Center, Missoula, Montana
  - CHI Health Saint Francis, Grand Island, Nebraska
  - CHI Health Good Samaritan, Kearney, Nebraska
  - Nebraska Cancer Specialists/Oncology Hematology West PC - MECC, Omaha, Nebraska
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Oncology Associates PC, Omaha, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Alegent Health Lakeside Hospital, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Summit Medical Group, Berkeley Heights, New Jersey
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - Summit Health - Florham Park Campus, Florham Park, New Jersey
  - The Cancer Institute of New Jersey Hamilton, Hamilton, New Jersey
  - Jersey City Medical Center, Jersey City, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Sidney Kimmel Cancer Center Washington Township, Sewell, New Jersey
  - Robert Wood Johnson University Hospital Somerset, Somerville, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - NYU Langone Hospital - Brooklyn, Brooklyn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Memorial Sloan Kettering Commack, Commack, New York
  - Glens Falls Hospital, Glens Falls, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - NYU Langone Hospital - Long Island, Mineola, New York
  - Mount Sinai Chelsea, New York, New York
  - Bellevue Hospital Center, New York, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - Mount Sinai West, New York, New York
  - Mount Sinai Hospital, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Rochester, Rochester, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York
  - Wilmot Cancer Institute at Webster, Webster, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Duke Women's Cancer Care Raleigh, Raleigh, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Essentia Health Cancer Center-South University Clinic, Fargo, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Essentia Health - Jamestown Clinic, Jamestown, North Dakota
  - OhioHealth O'Bleness Hospital, Athens, Ohio
  - UHHS-Chagrin Highlands Medical Center, Beachwood, Ohio
  - Geauga Hospital, Chardon, Ohio
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - Bethesda North Hospital, Cincinnati, Ohio
  - TriHealth Cancer Institute-Westside, Cincinnati, Ohio
  - TriHealth Cancer Institute-Anderson, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - Cleveland Clinic Cancer Center/Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Columbus Oncology and Hematology Associates Inc, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Delaware Health Center-Grady Cancer Center, Delaware, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Columbus Oncology and Hematology Associates, Dublin, Ohio
  - Dublin Methodist Hospital, Dublin, Ohio
  - OhioHealth Mansfield Hospital, Mansfield, Ohio
  - OhioHealth Marion General Hospital, Marion, Ohio
  - Hillcrest Hospital Cancer Center, Mayfield Heights, Ohio
  - UH Seidman Cancer Center at Lake Health Mentor Campus, Mentor, Ohio
  - OhioHealth Pickerington Methodist Hospital, Pickerington, Ohio
  - ProMedica Flower Hospital, Sylvania, Ohio
  - ProMedica Toledo Hospital/Russell J Ebeid Children's Hospital, Toledo, Ohio
  - OhioHealth Westerville Medical Campus/Westerville Cancer Center, Westerville, Ohio
  - UH Seidman Cancer Center at Saint John Medical Center, Westlake, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Mercy Hospital Oklahoma City, Oklahoma City, Oklahoma
  - Saint Alphonsus Cancer Care Center-Baker City, Baker City, Oregon
  - Saint Charles Health System, Bend, Oregon
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Bay Area Hospital, Coos Bay, Oregon
  - Providence Hood River Memorial Hospital, Hood River, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Saint Alphonsus Cancer Care Center-Ontario, Ontario, Oregon
  - Providence Willamette Falls Medical Center, Oregon City, Oregon
  - Legacy Good Samaritan Hospital and Medical Center, Portland, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Saint Charles Health System-Redmond, Redmond, Oregon
  - Legacy Meridian Park Hospital, Tualatin, Oregon
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Saint Luke's Cancer Center - Allentown, Allentown, Pennsylvania
  - Saint Luke's University Hospital-Bethlehem Campus, Bethlehem, Pennsylvania
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Christiana Care Health System-Concord Health Center, Chadds Ford, Pennsylvania
  - Chambersburg Hospital, Chambersburg, Pennsylvania
  - Pocono Medical Center, East Stroudsburg, Pennsylvania
  - Saint Luke's Hospital-Anderson Campus, Easton, Pennsylvania
  - Ephrata Cancer Center, Ephrata, Pennsylvania
  - Adams Cancer Center, Gettysburg, Pennsylvania
  - WellSpan Medical Oncology and Hematology, Hanover, Pennsylvania
  - Lehigh Valley Hospital-Hazleton, Hazleton, Pennsylvania
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - Sechler Family Cancer Center, Lebanon, Pennsylvania
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania
  - Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Jefferson Torresdale Hospital, Philadelphia, Pennsylvania
  - Saint Luke's Hospital - Upper Bucks Campus, Quakertown, Pennsylvania
  - Saint Luke's Hospital - Monroe Campus, Stroudsburg, Pennsylvania
  - Chester County Hospital, West Chester, Pennsylvania
  - Asplundh Cancer Pavilion, Willow Grove, Pennsylvania
  - WellSpan Health-York Cancer Center, York, Pennsylvania
  - WellSpan Health-York Hospital, York, Pennsylvania
  - Women and Infants Hospital, Providence, Rhode Island
  - Gibbs Cancer Center-Gaffney, Gaffney, South Carolina
  - Gibbs Cancer Center-Pelham, Greer, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - SMC Center for Hematology Oncology Union, Union, South Carolina
  - Avera Cancer Institute-Aberdeen, Aberdeen, South Dakota
  - Avera Cancer Institute - Mitchell, Mitchell, South Dakota
  - Avera Cancer Institute at Pierre, Pierre, South Dakota
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Avera Cancer Institute at Yankton, Yankton, South Dakota
  - Vanderbilt-Ingram Cancer Center at Franklin, Franklin, Tennessee
  - Vanderbilt-Ingram Cancer Center Cool Springs, Franklin, Tennessee
  - Vanderbilt Breast Center at One Hundred Oaks, Nashville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Parkland Memorial Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Fort Worth, Fort Worth, Texas
  - Houston Methodist Hospital, Houston, Texas
  - Memorial Hermann Texas Medical Center, Houston, Texas
  - Methodist Willowbrook Hospital, Houston, Texas
  - Houston Methodist West Hospital, Houston, Texas
  - Houston Methodist Saint John Hospital, Nassau Bay, Texas
  - UT Southwestern Clinical Center at Richardson/Plano, Richardson, Texas
  - Houston Methodist The Woodlands Hospital, The Woodlands, Texas
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - Providence Regional Cancer System-Aberdeen, Aberdeen, Washington
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Providence Regional Cancer System-Centralia, Centralia, Washington
  - Swedish Cancer Institute-Edmonds, Edmonds, Washington
  - Providence Regional Cancer Partnership, Everett, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - Providence Regional Cancer System-Lacey, Lacey, Washington
  - PeaceHealth Saint John Medical Center, Longview, Washington
  - Skagit Regional Health Cancer Care Center, Mount Vernon, Washington
  - Swedish Medical Center-Ballard Campus, Seattle, Washington
  - Fred Hutchinson Cancer Center, Seattle, Washington
  - Swedish Medical Center-Cherry Hill, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - University of Washington Medical Center - Montlake, Seattle, Washington
  - PeaceHealth United General Medical Center, Sedro-Woolley, Washington
  - Saint Michael Cancer Center, Silverdale, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - Cancer Care Northwest-Valley, Spokane, Washington
  - Cancer Care Northwest-North Spokane, Spokane, Washington
  - Legacy Salmon Creek Hospital, Vancouver, Washington
  - Providence Saint Mary Regional Cancer Center, Walla Walla, Washington
  - United Hospital Center, Bridgeport, West Virginia
  - WVUH-Berkely Medical Center, Martinsburg, West Virginia
  - West Virginia University Healthcare, Morgantown, West Virginia
  - Camden Clark Medical Center, Parkersburg, West Virginia
  - Princeton Community Hospital, Princeton, West Virginia
  - Wheeling Hospital/Schiffler Cancer Center, Wheeling, West Virginia
  - Duluth Clinic Ashland, Ashland, Wisconsin
  - Northwest Wisconsin Cancer Center, Ashland, Wisconsin
  - Aurora Cancer Care-Southern Lakes VLCC, Burlington, Wisconsin
  - Aurora Saint Luke's South Shore, Cudahy, Wisconsin
  - Aurora Health Care Germantown Health Center, Germantown, Wisconsin
  - Aurora Cancer Care-Grafton, Grafton, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Essentia Health-Hayward Clinic, Hayward, Wisconsin
  - Tamarack Health Hayward Medical Center, Hayward, Wisconsin
  - Aurora Cancer Care-Kenosha South, Kenosha, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Aurora Bay Area Medical Group-Marinette, Marinette, Wisconsin
  - Aurora Cancer Care-Milwaukee, Milwaukee, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - ProHealth D N Greenwald Center, Mukwonago, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - ProHealth Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - Saint Vincent Hospital Cancer Center at Oconto Falls, Oconto Falls, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Aurora Cancer Care-Racine, Racine, Wisconsin
  - Saint Vincent Hospital Cancer Center at Sheboygan, Sheboygan, Wisconsin
  - Sheboygan Physicians Group, Sheboygan, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Essentia Health-Spooner Clinic, Spooner, Wisconsin
  - Saint Vincent Hospital Cancer Center at Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Essentia Health Saint Mary's Hospital - Superior, Superior, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - ProHealth Waukesha Memorial Hospital, Waukesha, Wisconsin
  - UW Cancer Center at ProHealth Care, Waukesha, Wisconsin
  - Aurora Cancer Care-Milwaukee West, Wauwatosa, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
  - Memorial Hospital of Laramie County, Cheyenne, Wyoming
  - Billings Clinic-Cody, Cody, Wyoming
- Japan (11):
  - Tohoku University School of Medicine, Sendai, Aoba-ku
  - Ehime University Hospital, Tōon, Ehime
  - Kure Medical Center and Chugoku Cancer Center, Kure, Hiroshima
  - Hokkaido University Hospital, Sapporo, Hokkaido
  - Hyogo Cancer Center, Akashi, Hyōgo
  - Iwate Medical University Hospital, Shiwa-gun, Iwate
  - Kagoshima City Hospital, Kagoshima, Kagoshima-ken
  - The Cancer Institute Hospital Of JFCR, Koto-ku, Tokyo
  - Keio University, Shinjuku-ku, Tokyo
  - Jikei University School of Medicine, Minato-ku, Tokyo
  - Okayama University Hospital, Okayama
- Puerto Rico (7):
  - Cancer Center-Metro Medical Center Bayamon, Bayamón
  - Puerto Rico Hematology Oncology Group, Bayamón
  - Doctors Cancer Center, Manatí
  - San Juan Community Oncology Group, San Juan
  - Centro Comprensivo de Cancer de UPR, San Juan
  - PROncology, San Juan
  - San Juan City Hospital, San Juan